CLINICAL TRIAL: NCT05415540
Title: Changes in the Quality of Life and Experience of Young Women With Utero-vaginal Aplasia (MRKHPSY)
Brief Title: Evolution of the Quality of Life and Experience of Young Women With Utero-vaginal Aplasia (MRKHPSY)
Acronym: MRKHPSY
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Foundation for Rare Diseases (Unknown); Necker Imagine Foundation (Unknown); Laboratory of Clinical Psychology, Psychopathology and Psychoanalysis (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211596; 2021-A02881-40 (Other: ID-RCB Number)
Record Dates: First submitted 2022-05-02; First posted 2022-06-13 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Mrkh Syndrome
Keywords: Mayer-Rokitansky-Kuster-Hauser Syndrome; Quality of life; Utero-vaginal aplasia
MeSH Terms: conditions — Mullerian aplasia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires — Subjects included in the study will answer questionnaires

SUMMARY:
This study aims to evaluate the global evolution of the quality of life on patients diagnosed with MRKH syndrome (Mayer-Rokitansky-Kuster-Hauser), 8 to 10 years after the first research.

DETAILED DESCRIPTION:
Between 2012 and 2015, the French national reference center for rare gynecological pathologies (PGR) has conducted a study with 2 axis: a medical and a psychological section (clinical trial number NCT01911884).

The medical axis's aim was to compare the global and sexual quality of life of MRKH patients according to the mode of care (surgical or non-surgical) for vaginal aplasia. A total of 131 patients, with a mean age of 26.5 (±5.5) years old, were recruited for the study.

The quality of life was assessed considering 3 quality of life scales: global (WHOQOL-BREF) and sexual (FSFI and FSDS-R).

Quality of life scores and vaginal depth were compared and revealed that the surgery was not superior to self-dilation, whether in terms of quality of life or anatomical results. In addition, surgery was associated with complications in half of the cases. It should be mentioned that the overall quality of life of all 131 patients was similar to that of the general population, but significantly impaired in the psychosocial dimension in the younger patients. Notably, the quality of sexual life was not impaired with FSFI scores similar to those of the general population, but there was a profound sexual distress in nearly 71% of patients according to FSDS-R scores.

The psychological component of this initial research (called T1) focused specifically on the psychological, and more widely on the psychosocial, impact of the diagnosis of utero-vaginal aplasia in adolescent girls. 40 patients out of the 131 in the medical component participated (the first 40 contacted to participate in the medical component research). The results revealed a real experience of disability, and unexpectedly, addictive reactionary disorders (anorexia/bulimia or sport addiction), and an overrepresentation of heterosexual orientation compared to the general population. The absence of a uterus led to severe moral suffering regarding projections of access to biological motherhood.

This new research (called T2) involves the same population as T1 with the object of making each patient her own witness.

The purpose of the current study is to assess the evolution of this suffering, 8 to 10 years after the T1 study, using the same methodology as the previous study. The investigators hope to find an improvement in quality of life, a disappearance of addictive disorders and possibly a more vivid, but painful expression due to age, of the desire for motherhood, even if the uterus transplant is a source of hope.

Finding predictive factors of psychosocial difficulties would allow teh investigators to improve care practices, mainly psychological, which could also benefit other women with a rare disease affecting their sexuality and/or fertility.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged of 18 years old or older
* Patient who participated in the initial T1 psychological component of the previous study (MRKH protocol)

Exclusion Criteria

- Refusal to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patient who participated in the initial T1 psychological component of the previous study (MRKH protocol)
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Evaluation of global quality of life | Day 0
  Evaluated by the World Health Organization Quality Of Life Brief Version (WHOQOL-BREF)

SECONDARY OUTCOMES:
Socio-professional integration | Day 0
  Socio-professional integration based on professional integration criteria. The potential consequences of this malformation on socio-professional integration are also diagnosed during the semi-directive clinical consultation and with the quality of life scale:
  - Total score WHOQOL-BREF
Socio-professional integration | Day 0
  Socio-professional integration based on professional integration criteria. The potential consequences of this malformation on socio-professional integration are also diagnosed during the semi-directive clinical consultation and with the quality of life scale:
  - item 18 score (How satisfied are you with your capacity for work?)
Socio-professional integration | Day 0
  Socio-professional integration based on professional integration criteria. The potential consequences of this malformation on socio-professional integration are also diagnosed during the semi-directive clinical consultation and with the quality of life scale:
  -qualitative components mentioned during the clinical consultation regarding education and socio-professional integration
Sexual quality of life | Day 0
  Sexual quality of life is assessed by two sex life self-questionnaires (Female Sexual Function Index FSFI and Female Sexual Dysfunction Scale-Revised FSFD).
Addictive behavioural disorders | Day 0
  Description : Addictive behavioural disorders are diagnosed during the semi-directive clinical consultation. The semi-directive clinical consultation aims to promote the production of a speech by the patient on a given theme. This will be about the evolution of the personal history when the diagnosis was announced and the medical and/or surgical consequences that this diagnosis induced.
Desire for motherhood | Day 0
  The desire for motherhood is identified during the semi-directive clinical consultation.
The modalities to access to maternity | Day 0
  The modalities to access to maternity is identified during the semi-directive clinical consultation with three items: adoption, surrogacy, uterus transplantation;
Modalities of their psychic functioning | Day 0
  by the semi-directive clinical interview and the Rorschach&TAT with 13 variables:
  * Adaptation to reality
  * Type of anxiety:castration, loss of object, fragmentation, intrusion
  * Body image and characteristics of human responses :whole, partial, blurred, attacked
  * Self-representation:solid/fragile
  * Capacity to deploy conflictual scenarios
  * Female identification capability
  * Access to ambivalence
  * Modalities of thought investment: quality of laboration of the modes of apprehension: good/inadequate
  * Quality of psychic functioning and defensive range: flexible and adapted/rigid and adapted/flexible and inadapted/rigid and inadapted

CONTACTS AND LOCATIONS:
Overall Officials: Alaa CHEIKHELARD, Doctor, Principal Investigator; Karinne Gueniche, MD, PhD, Study Director
Locations (1):
- Necker Children's Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No